CLINICAL TRIAL: NCT02107872
Title: Study to Assess the Safety and Tolerability of Multiple Ascending Doses of REGN1500
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1500-CL-1321
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Metabolic Disorders
MeSH Terms: conditions — Metabolic Diseases | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- dosing cohort 1 (Experimental): Patients will receive REGN1500 or placebo in dosing cohort 1
  Interventions: Drug: REGN1500; Drug: placebo
- dosing cohort 2 (Experimental): Patients will receive REGN1500 or placebo in dosing cohort 2
  Interventions: Drug: REGN1500; Drug: placebo
- dosing cohort 3 (Experimental): Patients will receive REGN1500 or placebo in dosing cohort 3
  Interventions: Drug: REGN1500; Drug: placebo
- dosing cohort 4 (Experimental): Patients will receive REGN1500 or placebo in dosing cohort 4
  Interventions: Drug: REGN1500; Drug: placebo
- dosing cohort 5 (Experimental): Patients will receive REGN1500 or placebo in dosing cohort 5
  Interventions: Drug: REGN1500; Drug: placebo

INTERVENTIONS:
Drug: REGN1500
Drug: placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, multiple ascending dose study to assess the safety, tolerability, pharmacokinetic (PK), immunogenicity, and pharmacodynamic (PD) effects of REGN1500 in patients with a metabolic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent
* Otherwise healthy men and women ages 18 to 65 years, inclusive
* Body mass index of 18.0 kg/m2to 38.0 kg/m2, inclusive
* Normal standard 12-lead ECG
* Willing to refrain from the consumption of alcohol for 24 hours prior to each study visit
* Willing to consistently maintain his/her usual diet for the duration of the study
* Willing to refrain from strenuous exercise for the duration of the trial
* Willing and able to comply with clinic visits and study-related procedures
* For sexually active men and women of childbearing potential, willingness to utilize adequate contraception and not become pregnant (or have their partner[s] become pregnant) during the full duration of the study.

Exclusion Criteria:

* Any clinically significant abnormalities observed during the screening visit
* History of drug or alcohol abuse within 1 year of screening
* Receipt of another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit.
* Significant concomitant illness or history of significant illness such as cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease, or any other illness or condition that may adversely affect the subjects participation in this study
* Known history of human immunodeficiency virus (HIV) antibody; and/or positive hepatitis B surface antigen (HBsAg), and/or positive hepatitis C antibody (HCV) at the screening visit
* Hospitalization for any reason within 60 days of screening
* History or presence of malignancy within 5 years prior to the screening visit (other than successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma, and/or localized carcinoma in situ of the cervix
* Any medical or psychiatric condition which, in the opinion of the investigator, would place the subject at risk, interfere with participation in the study or interfere with the interpretation of the study results
* Any subject who is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff directly involved in the conduct of the protocol, or family member of staff involved in the conduct of the protocol
* Pregnant or breast-feeding women

Note: The information listed above is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial and not all inclusion/ exclusion criteria are listed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety | visit 1 to day 183 (EOS)
  Safety of REGN1500 will be assessed by physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory evaluations from visit 1 to day 183 [EOS (end of study)]

SECONDARY OUTCOMES:
Serum concentration | visit 1 to day 183
  Serum concentration, amount of REGN1500 in the circulation, over time (visit 1 to day 183)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- United States (4):
  - Daytona Beach, Florida
  - Evansville, Indiana
  - Dallas, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Ahmad Z, Banerjee P, Hamon S, Chan KC, Bouzelmat A, Sasiela WJ, Pordy R, Mellis S, Dansky H, Gipe DA, Dunbar RL. Inhibition of Angiopoietin-Like Protein 3 With a Monoclonal Antibody Reduces Triglycerides in Hypertriglyceridemia. Circulation. 2019 Aug 6;140(6):470-486. doi: 10.1161/CIRCULATIONAHA.118.039107. Epub 2019 Jun 27. PMID 31242752